CLINICAL TRIAL: NCT04079868
Title: Models of Primary Osteoporosis Screening in Male Veterans
Acronym: MOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IIR 17-202
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Osteoporosis; Osteopenia; Osteoporotic Fracture
Keywords: Osteoporosis; Osteopenia; Osteoporotic fracture; Age-Related Osteoporosis; Bone Loss, Age-Related
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Osteoporotic Fractures

STUDY DESIGN:
Intervention Model Description: Stratified, block randomization will be used. A statistician unaware of team identity will randomize PACTs in blocks of 2 within strata to ensure similar distributions. If insufficient numbers of PACTs are recruited within small CBOCs, they will be combined with other similar CBOCs (rural vs. urban) for randomization.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked to the group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bone Health Service arm (Experimental): Interventional arm
  Interventions: Behavioral: Bone Health Service Model
- Usual care (control) arm (No Intervention): This arm represents a "no practice management support" control group.

INTERVENTIONS:
Behavioral: Bone Health Service Model — Patients in PACTs randomized to the BHS model will have osteoporosis screening, education, and follow-up handled centrally by the bone health team.
  Arms: Bone Health Service arm

SUMMARY:
Models of Osteoporosis Screening in Male Veterans aims to test 1 distinct care model of primary osteoporosis screening in men within the VA healthcare setting. All care models deliver VA recommended osteoporosis screening and treatment to high-risk Veterans by appropriate Durham VA clinical staff. The MOPS project will evaluate patient, provider and facility outcomes to determine the effectiveness of each intervention.

DETAILED DESCRIPTION:
Background/Purpose:

Osteoporosis is under-recognized in older men. At age 50 years, 1 in 5 men can expect to suffer a major osteoporotic fracture in their remaining lifetime, comparable to the risk of prostate cancer. Men are more than twice as likely as women to experience complications after a fracture, and have greater excess mortality after hip fracture. Because risk factors are common in Veterans, osteoporosis is particularly prevalent in the Veterans Health Administration (VA) system. More than half of male Veterans over age 50 years have osteopenia or osteoporosis, a rate nearly double the non-Veteran population.

Fractures resulting from osteoporosis have negative consequences on functional status, mortality, and quality of life, with high rates of pain, depression, and loss of independence. After a hip fracture, nearly 75% of patients spend time in a nursing facility, and only 20% regain their prior level of ambulation. Many fractures are associated with substantial excess mortality; men with a hip fracture have excess annual mortality of 20% that persists up to 10 years. Osteoporotic fractures also have an important economic impact. It is estimated that hip fractures result in 43 million dollars of excess cost to the VHA annually.

Osteoporosis screening and treatment services within VA are ineffective overall. Overall, screening rates were 8% for men over age 65; far lower than expected based on the prevalence of osteoporosis risk factors in the population. Moreover, even among men in whom screening was completed, it was not associated with lower overall fracture rates because osteoporosis treatment and adherence following screening were extremely low.

Attempts to improve osteoporosis screening using traditional quality improvement programs have been minimally effective. Electronic health record (EHR) alerts alone do not improve osteoporosis screening rates and do nothing to address adherence. However, one distinct osteoporosis screening paradigm has been suggested, and form the scientific premise for the models proposed in this application. A fracture Liaison Service (referred to here as "Bone Health Service", BHS) represents a centralized model that has been successful in improving secondary osteoporosis screening and treatment adherence after a fracture has already occurred. In this model, a team of nurses led by a bone specialist identify patients with fracture within the entire health system, and arrange for evaluation and treatment. Such models have reduced 2-year fracture rates by 56% and are cost saving or highly cost-effective.

Objectives:

The investigators propose a pragmatic group randomized trial of PACT teams from both Durham and Richmond VAMC's. A PACT's will be randomized into 2 groups: a control group (no additional support), and a centralized Bone Health Service (BHS) model where teams will manage the screening and treatment of high-risk for fracture male Veterans.

Outcomes for all patients eligible for osteoporosis screening within the randomized PACTs will be assessed by investigators masked to group assignment. Outcomes for PACT providers will be assessed using qualitative methods (nominal group technique).

Patient-level outcomes:

* Eligible proportion screened
* Medication adherence
* PACT fracture rates
* Harms
* Bone mineral density

Provider and facility level outcomes:

* Change in Dual-energy X-ray absorptiometry (DXA) volume
* Bone mineral density (sub-sample of patients)
* Change in metabolic bone disease clinic volume
* PACT provider time and satisfaction (qualitative analyses)

Health system and policy level outcomes

* Program cost effectiveness

Methodology:

The investigators will compare the 1 screening models by enrolling, screening and randomizing PACT teams. 39 teams will be randomized, an estimated 24 teams at the Durham VA health care system and 15 at the Richmond VA medical center. Teams will be randomized to 1 of 2 arms: Bone Health Service or usual care (no additional support). A sub-set of providers will be recruited to complete a nominal group qualitative interview during year 3. Also a random sub-set of patients (900) will be recruited to complete a DXA scan to measure bone density beginning in year 4. Outcomes will be assessed at year 1, 2, 3, and 4.

ELIGIBILITY:
Inclusion Criteria:

PACT Team inclusion criteria:

* Provider with at least 0.75 FTE
* Provider has completed training (i.e., PACT teams led by residents and fellows are excluded)
* Care for male Veterans >65 years (i.e., Women's Health PACTs are excluded)

Patient Inclusion criteria:

* No prior fracture or osteoporosis diagnosis
* At least 1 VA Undersecretary Guideline risk factor (weight loss >20% in 5 years; BMI <25 kg/m2; diabetes; pernicious anemia; gastrectomy; anticonvulsants; glucocorticoids; androgen deprivation therapy; hyperthyroidism; hyperparathyroidism; rheumatoid arthritis; alcohol dependence; chronic lung disease; chronic liver disease; stroke; Parkinsonism; prostate cancer; and current smoking).

Patients (enrolled in year 4/5 sub-sample) inclusion criteria:

* Men aged 65-85 years
* Enrolled in eligible PACT team for at least 2 years
* Meet 1 or more criteria for osteoporosis screening as the protocol at PACT enrollment.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3512 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen S Colon-Emeric, MD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (3):
- United States (3):
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colon-Emeric C, Lee R, Lyles KW, Zullig LL, Sloane R, Pieper CF, Nelson RE, Adler RA. Remote Bone Health Service for Osteoporosis Screening in High-Risk Men: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2025 Oct 1;185(10):1218-1224. doi: 10.1001/jamainternmed.2025.4150. PMID 40853653

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Primary care teams
Period: Overall Study
Arm/Group | Bone Health Service Arm | Usual Care (Control) Arm
Started | 1888; 20 Primary care teams | 1624; 19 Primary care teams
Completed | 1688; 18 Primary care teams | 1424; 17 Primary care teams
Not Completed | 200; 2 Primary care teams | 200; 2 Primary care teams
Not completed — Lost to Follow-up | 100 | 200
Not completed — Physician Decision | 100 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bone Health Service Arm | Usual Care (Control) Arm | Total
Number analyzed (Participants) | 1688 | 1424 | 3112
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (5.2) | 73.8 (5.4) | 73.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1688 | 1424 | 3112
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 695 | 565 | 1260
  White | 930 | 818 | 1748
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 63 | 41 | 104

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Screened for Osteoporosis
Description: Proportion of men who received DXA screening for for osteoporosis. Numerator is the number of men with a completed screening DXA, denominator is all patients meeting current osteoporosis screening criteria
Time Frame: through study completion, an average of 1.5 years
Measure: Number; unit: participants
Arm/Group | Bone Health Service Arm | Usual Care (Control) Arm
Number analyzed (Participants) | 1688 | 1424
participants | 830 | 33

2. Primary Outcome: Bone Mineral Density T-score at the Femoral Neck
Description: Bone mineral density in gm/cm2 as measured by DXA, converted to T-score by the densitometer manufacturer. The T score reflects the number of standard deviations away from the mean bone density of young healthy women as defined in the National Health and Nutrition Survey. Lower T-scores reflect worse bone density, and T-scores <= -1 are consistent with osteopenia or osteoporosis. This outcome was measured in a random subset of enrolled patients (target n=25 per primary care team), regardless of whether or not they had undergone osteoporosis screening during the study period.
Time Frame: 2 years after the primary care team's start date
Measure: Mean (Standard Deviation); unit: T score femoral neck
Arm/Group | Bone Health Service Arm | Usual Care (Control) Arm
Number analyzed (Participants) | 413 | 353
T score femoral neck | -0.55 (1.28) | -0.70 (1.25)

3. Secondary Outcome: Gastrointestinal Medication Prescriptions
Description: This is a measure of potential harm from osteoporosis treatment. Numerator is number of men with new prescription for proton pump inhibitor or H2 blocker, denominator is all men eligible for osteoporosis screening
Time Frame: through study completion, an average of 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Health Service Arm | Usual Care (Control) Arm
Number analyzed (Participants) | 1688 | 1424
Participants | 562 | 473

4. Secondary Outcome: Osteoporosis Medication Adherence (Proportion of Days Covered)
Description: For patients started on osteoporosis medications, numerator is the total number of dispensed units, denominator is the number of days between the first medication prescription and medication discontinuation, death, or end of the study period
Time Frame: through study completion, an average of 1.5 years
Measure: Mean (Standard Deviation); unit: proportion of days covered by meds
Arm/Group | Bone Health Service Arm | Usual Care (Control) Arm
Number analyzed (Participants) | 113 | 4
proportion of days covered by meds | 0.92 (0.24) | 1.0 (0.13)

5. Secondary Outcome: Proportion of Patients Initiating Osteoporosis Medication (%)
Description: Numerator is number of patients prescribed osteoporosis medications, denominator is number of patients eligible for osteoporosis medications based on their DXA results
Time Frame: through study completion, an average of 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Health Service Arm | Usual Care (Control) Arm
Number analyzed (Participants) | 137 | 9
Participants | 113 | 4

6. Secondary Outcome: Osteoporosis Medication Persistence (Days)
Description: Among participants who were prescribed an osteoporosis medication, the mean number of days between the first dispensing date until a gap in medication prescription of >=90 days occurred
Time Frame: through study completion, up to 2 years
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bone Health Service Arm | Usual Care (Control) Arm
Number analyzed (Participants) | 113 | 4
days | 657 (366) | 730 (480)

7. Secondary Outcome: Proportion With Fractures
Description: Numerator is number of men with a confirmed fracture during study follow-up, denominator is all men eligible for osteoporosis screening at baseline
Time Frame: through study completion, an average of 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Health Service Arm | Usual Care (Control) Arm
Number analyzed (Participants) | 1688 | 1424
Participants | 31 | 29

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Bone Health Service Arm | Usual Care (Control) Arm
All-Cause Mortality (participants affected / at risk) | 135/1688 | 89/1424
Serious Adverse Events (participants affected / at risk) | 0/1688 | 0/1424
Other Adverse Events (participants affected / at risk) | 1/1688 | 0/1424
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bone Health Service Arm (N=1688) | Usual Care (Control) Arm (N=1424)
Drug interaction (Endocrine disorders) | 1 | 0 — Interaction between calcium supplements prescribed in BHS patient with prescribed levothyroxine with asymptomatic TSH elevation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT04079868/Prot_001.pdf
  • Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT04079868/SAP_002.pdf
  • Informed Consent Form (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT04079868/ICF_000.pdf